CLINICAL TRIAL: NCT01696331
Title: Impact of Text Messaging on Adherence in Adolescent Liver Transplant Patients
Brief Title: Text Messaging for Adherence in Adolescent Liver Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rebecca Berquist McKenzie, Clinical Instructor, Department of Pediatric Gastroenterology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25318
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Liver Transplant; Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Text Message Reminder (Experimental)
  Interventions: Behavioral: Text Message Reminder

INTERVENTIONS:
Behavioral: Text Message Reminder — Sent TM reminder at beginning and end of each month that corresponded to required lab frequency. Patients were able to send autoresponses.

SUMMARY:
Text message reminders will improve adherence to lab tests in adolescent liver transplant recipients.

DETAILED DESCRIPTION:
Adolescent patients who received a liver transplant will be recruited to participate in receiving text message reminders for lab tests. They will be send de-identified messages according to their required lab schedule. The investigators will monitor their adherence to lab tests as well as medication and clinic visits. They will also have a questionnaire about their medical regimen before and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient >12 years
* Received liver transplant
* Followed by Stanford Liver Transplant Team

Exclusion Criteria:

* No personal cell phone

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Adherence to lab tests | One year

SECONDARY OUTCOMES:
Texting responses | 1 year
  Correspondence between actual completion of tests versus reported

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States